CLINICAL TRIAL: NCT01649609
Title: Using mTOR Inhibitors in the Prevention of BK Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Pfizer (Industry); Cornell University (Other)
Responsible Party: Principal Investigator, Sumit Mohan, MD, Assistant Professor of Clinical Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAI9004; WS2036051 (Other: Pfizer)
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: BK Viremia; BK Nephropathy
Keywords: BK Viremia; BK Nephropathy; mTOR inhibitor; renal transplant
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduction of standard immunosuppression (Active Comparator): Low dose Tacrolimus with low dose Mycophenolate acid
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate acid
- mTOR Arm (Active Comparator): Low dose Sirolimus with low dose Mycophenolate acid (mTOR Substitution)
  Interventions: Drug: Mycophenolate acid; Drug: Sirolimus

INTERVENTIONS:
Drug: Tacrolimus — Reduction of standard immunosuppression - The standard of care immunosuppression treatment commonly used for renal transplant patients
  Other Names: Prograf
  Arms: Reduction of standard immunosuppression
Drug: Mycophenolate acid — Myfortic or CellCept - The standard of care immunosuppression treatment most commonly used for renal transplant patients
  Other Names: mycophenolate antimetabolite
Drug: Sirolimus — mTOR Substitution - Replacing tacrolimus (a calcineurin inhibitor) with sirolimus (an mTOR inhibitor) along with reduction of mycophenolic acid
  Other Names: Rapamune
  Arms: mTOR Arm

SUMMARY:
BK virus infections after kidney transplant are increasing and can result in damage to the transplanted kidney. Currently, the universally accepted treatment is to decrease the strength of the antirejection medications but it is unclear what medications should be lowered and to what extent. The investigators propose to perform a study with patients who have BK virus detected in their blood during routine screening that appears to be increasing. The investigators will use two different strategies that involve different combinations of standard anti-rejection medications at lower dosages. Patients will be assigned to one of the two groups in a random manner across the two hospitals participating in the study. Patients will be followed for at least a year to determine if one strategy was more effective than the other in preventing an increase in the number of viruses in the blood stream and whether either one was more effective in reducing the negative impact of the infection on the functioning of the transplanted kidney.

DETAILED DESCRIPTION:
The incidence of BK viremia, an early complication after renal transplantation and the associated rates of graft loss resulting from BK nephropathy have been steadily rising since a series of cases that were reported in the mid-1990's. While this is at least partly related to the introduction of newer immunosuppressive agents, recent United Network for Organ Sharing (UNOS) data analyses suggest that there is a continuing rise in the incidence of BK viremia and associated nephropathy with a 3.5% incidence rate in 2009 representing a dramatic rise from just 0.9% only 4 years earlier. Single center data reports have suggested much lower rates of BK viremia and nephropathy in cohorts treated with mTOR (mammalian target of rapamycin) based immunosuppressive regimens when compared to the overall national incidence rates. Recent data has demonstrated that calcineurin inhibitors at concentrations routinely used in clinical practice interfere with the BK virus specific T cell responses; an interference that is not seen to occur with mTOR inhibitors. Further, recent evidence that inhibition of the mTOR pathway has a direct and consequential negative impact on BK infected cells provides additional insight into the observed benefit associated with mTOR inhibitors. The growing problem of BK viremia among renal transplant patients is further compounded by the absence of effective management strategies that have been tested in a rigorous or controlled setting - a fact that was highlighted in a recent systematic review. The cornerstone for management so far has been the reduction of immunosuppression, largely based on the outcome of a single center study of screening patients for viremia and following with preemptive lowering of immunosuppression. Conversion from calcineurin inhibitors to mTOR inhibitors has been reported in small case series to be an effective measure that appears to be superior to merely lowering immunosuppression; however, this approach has not been tested with a robust clinical study design.

Currently, the diagnosis of BK nephropathy requires a renal biopsy, an invasive procedure with its own risks. In addition, identification of patients with viremia who progress to nephropathy and subsequent graft failure i.e. prognostication does not appear possible with the renal biopsy results at present. Validation of potential non-invasive biomarkers provides a unique opportunity for both detection and risk stratification of patients with BK viremia subsequent failure, which could lead to more informed therapeutic interventions while supporting the development of newer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients age 18 years or over

Exclusion Criteria:

* Patients with multiorgan transplants
* Patients on immunosuppressive regimens that include steroids or Sirolimus at the time of detection of viremia
* ABO incompatible renal transplants
* Three or more previous renal transplants
* Patients with contraindications to tacrolimus, sirolimus, mycophenolate mofetil or mycophenolic acid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Mohan, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Immunosuppression Reduction Arm: Those in the standard immunosuppression reduction arm experienced a reduction of the calcineurin inhibitor (i.e. tacrolimus) dosage to a goal level of 4-8 μg/L and reduction of the antimetabolite agent (mycophenolic acid/mycophenolate mofetil) to 50% of dose at the time of detection of viremia (once BK viremia PCR >5000 copies/mL).
- mTOR Substitution Arm: Those in the mTOR substitution arm experienced replacement of the calcineurin inhibitor (i.e. tacrolimus) with the mTOR agent, Sirolimus for a level of 6-10 μg/L coupled with reduction of the antimetabolite dose to 50% of the dose at the time of detection of the viremia (once BK viremia PCR >5000 copies/mL).
Period: Overall Study
Arm/Group | Standard Immunosuppression Reduction Arm | mTOR Substitution Arm
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Immunosuppression Reduction Arm | mTOR Substitution Arm | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 18 | 28
  >=65 years | 10 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.04 (14.12) | 52.39 (12.69) | 56.7 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 15 | 18 | 33
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 6 | 9
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Delayed Graft Function [Count of Participants; unit: Participants] | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With BK Viral Load <600 Copies/mL
Description: A Viral load of <600 copies/mL for at least 3 months indicates sustained clearance of BK viremia, confirmed by blood test
Time Frame: Up to 12 months from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Immunosuppression Reduction Arm | mTOR Substitution Arm
Number analyzed (Participants) | 20 | 20
Participants | 13 | 17

2. Secondary Outcome: Number of Participants With Incidence of BK Nephropathy
Description: The number of people with incidence of BK Nephropathy in each of the two Arms
Time Frame: Up to 24 months from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Immunosuppression Reduction Arm | mTOR Substitution Arm
Number analyzed (Participants) | 20 | 20
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: Up to 24 months
Arm/Group | Standard Immunosuppression Reduction Arm | mTOR Substitution Arm
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Immunosuppression Reduction Arm (N=20) | mTOR Substitution Arm (N=20)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) — Proteinuria > 1 gram
Rapa Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Pneumonitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes